CLINICAL TRIAL: NCT02396641
Title: Implementation of Consensus-based Standards for Best Supportive Care in a Clinical Trial: a Pilot Study
Brief Title: PCRC Best Supportive Care (PCRC BSC)
Acronym: PCRC BSC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Palliative Care Research Cooperative Group (Network); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); American Cancer Society, Inc. (Other); University of California, San Francisco (Other); Northwestern University (Other); University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00060650
Record Dates: First submitted 2015-03-18; First posted 2015-03-24 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2015-12

CONDITIONS: Feasibility of Best Supportive Care Delivery
Keywords: Best Supportive Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Study Arm (Experimental): This study arm consists of providers who will identify their baseline in Best Supportive Care, then have the intervention of using a Best Supportive Care checklist.
  Interventions: Other: Best Supportive Care Checklist

INTERVENTIONS:
Other: Best Supportive Care Checklist

SUMMARY:
The primary objective of this study is to formalize the delivery of BSC in advanced cancer trials. The first aim (to develop expert-derived consensus statements regarding components of supportive care in cancer clinical trials) and the second aim (to compare the extent to which documentation of current supportive care delivery in trials compares to the consensus statements) have been completed. The final aim of this study is to test the feasibility of thorough documentation of BSC delivery. That work is proposed as the primary aim of this study.

DETAILED DESCRIPTION:
Many cancer clinical trials are designed to evaluate the benefits of experimental anticancer drugs against best supportive care (BSC); many drugs have been registered based on very modest survival advantages when compared with BSC.

Universally across these studies, however, BSC control arms have not been standardized across sites in the way that trialists strive to standardize other interventions in clinical trials; are not consistent with contemporary palliative care practice; are not based on the extensive best available evidence; and are not described in any detail in most cases and certainly not sufficient detail to reproduce in subsequent studies. When reporting of BSC in trials is incomplete, the resulting data have uncertain internal and external validity.

Such poorly defined interventions and variation between sites is unacceptable for other aspects of a clinical trial. Furthermore, a poorly delivered BSC arm might systematically overestimate the performance of the intervention arm(s) in the study leading to poor decision making by clinicians and funders. With mounting evidence that early use of supportive/palliative care can improve patient outcomes, incomplete delivery of BSC might deprive patients of considerable benefit, potentially in the setting of far less toxicity.

In line with the CONSORT statement on reporting of clinical trials, our proposed study would seek to generate consensus-based standards for BSC definition (allowing this to be updated as new evidence becomes available), operationalize and measure outcomes in a clinical trial setting. In doing so, we intend to demonstrate: 1) the feasibility of thorough documentation of BSC, its delivery and measurement in a clinical trial; and 2) improved quality of life over standardized BSC. Specifically in terms of PCEOL research objectives, this study will develop an intervention designed to mitigate adverse physical and psychological symptoms and outcomes that focus especially on the beginning of the end-of-life phase.

This will be a prospective, single arm before and after consecutive cohort study of oncologists and patients. Initially, individual and institutional best practice in terms of supportive/palliative care delivery will be recorded across all sites (control period). Two months into study initiation, patients will complete pre-intervention patient ESAS and PNPC-sv assessment to measure their baseline care experience. At that point, all sites will simultaneously switch to the behavioral modification intervention (BSC checklist; experimental period). From that time forward, documentation of supportive care delivery will be documented via the BSC checklist and medical record review. At month four, physician acceptability and patient experience will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Must have incurable cancer
* A shortened life expectancy such that the treating clinician would not be surprised if the patient passed away within 6 months
* Karnofsky score ≥50
* Must be receiving anticancer therapy (including chemotherapy or hormonal therapy)
* By their clinician's best estimate, must be expected to receive at least two months of palliative anticancer therapy at the time of enrollment
* Must be under active management for cancer- or treatment-related symptoms.

Exclusion Criteria:

* Non-English speaking
* Unable to read or write
* Unable to travel to clinic for an appointment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Feasibility of thorough documentation of BSC delivery, consistent with BSC consensus statements, via the BSC checklist | 60 days

REFERENCES:
- [Result] Nipp RD, Currow DC, Cherny NI, Strasser F, Abernethy AP, Zafar SY. Best supportive care in clinical trials: review of the inconsistency in control arm design. Br J Cancer. 2015 Jun 30;113(1):6-11. doi: 10.1038/bjc.2015.192. Epub 2015 Jun 11. PMID 26068397
- [Result] Cherny NI, Abernethy AP, Strasser F, Sapir R, Currow D, Zafar SY. Improving the methodologic and ethical validity of best supportive care studies in oncology: lessons from a systematic review. J Clin Oncol. 2009 Nov 10;27(32):5476-86. doi: 10.1200/JCO.2009.21.9592. Epub 2009 Jun 29. PMID 19564538
- [Result] Zafar SY, Currow DC, Cherny N, Strasser F, Fowler R, Abernethy AP. Consensus-based standards for best supportive care in clinical trials in advanced cancer. Lancet Oncol. 2012 Feb;13(2):e77-82. doi: 10.1016/S1470-2045(11)70215-7. PMID 22300862
- [Result] Currow DC, Foley K, Zafar SY, Wheeler JL, Abernethy AP. The need for a re-evaluation of best supportive care studies reported to date. Br J Cancer. 2011 Feb 1;104(3):390-1. doi: 10.1038/sj.bjc.6606081. No abstract available. PMID 21285970